CLINICAL TRIAL: NCT00001560
Title: Clinical, Laboratory and Epidemiologic Pilot Studies of Individuals at High Risk for Viral-Associated Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970028; 97-C-0028; NCT00556582 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Acquired Immunodeficiency Syndrome; Kaposi's Sarcoma; Leukemia; Lymphoma; Tumor Virus Infection; HIV Infections
Keywords: AIDS; Multidisciplinary; Leukemia; Lymphoma; Kaposi's Sarcoma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sarcoma, Kaposi; Leukemia; Lymphoma; Tumor Virus Infections; HIV Infections

SUMMARY:
This protocol presents the rationale, 25-year historical review, and methods for multidisciplinary, low-risk studies of individuals referred to the NCI Viral Epidemiology Branch (VEB). Referrals are generally for unusual types of cancer or related conditions, known, or suspected to be related to viruses. Kaposi's sarcoma in two homosexual men evaluated in 1981 is a classic example. These referral cases provide the basis for pilot studies that generate hypotheses, the development of protocols for formal investigations of promising leads, and help to set priorities for VEB.

A VEB investigator who is a Staff Member at the NIH Clinical Center, interviews each subject, performs a physical examination, draws a blood sample, and, when appropriate for the disease or virus under study, obtains other clinically indicated biological specimens, such as urine, sputum, saliva, tears, semen, Pap smear, or cervical, anal, oral, or nasal swabs. On occasion, other relatively non-invasive studies may be indicated. Skin testing with conventional, licensed antigens for assessment of cellular immunity may be performed, and skin lesions may be biopsied or excised. Tumor or other tissue biopsies may be obtained when biopsy or surgery is clinically indicated for other reasons. Otherwise no surgery is performed, and no therapy is administered. Clinical referral to other components of NCI, NIH, or the private sector are made as needed. The biological specimens are frozen or otherwise preserved to be batch tested in current assays or future assays that will be developed. Such laboratory testing is performed either at VEB's own support laboratory, or collaboratively in other NCI, NIH, or extramural laboratories that have the needed expertise for the disease or virus under study.

Occasionally, repeated or more long-term evaluation is required. More often, a single evaluation in the NIH outpatient clinic, or either at a collaborating physician's office or other suitable site in the field, is sufficient. The VEB investigator provides counseling relevant to the virus or disease under study, and about the interim study results. He or she makes appropriate referral if needed (e.g., to the Genetic Epidemiology Branch for genetic counseling). Clinically relevant results and the VEB investigator's interpretation of these results, are provided in writing to the subject's primary caregiver. Confidentially of the information that is obtained is carefully protected. The results of the study are summarized for publication in the peer review literature.

DETAILED DESCRIPTION:
This protocol presents the rationale, 25-year historical review, and methods for multidisciplinary, low-risk studies of individuals referred to the NCI Viral Epidemiology Branch (VEB). Referrals are generally for unusual types of cancer or related conditions, known, or suspected to be related to viruses. Kaposi's sarcoma in two homosexual men evaluated in 1981 is a classic example. These referral cases provide the basis for pilot studies that generate hypotheses, the development of protocols for formal investigations of promising leads, and help to set priorities for VEB.

A VEB investigator who is a Staff Member at the NIH Clinical Center, interviews each subject, performs a physical examination, draws a blood sample, and, when appropriate for the disease or virus under study, obtains other clinically indicated biological specimens, such as urine, sputum, saliva, tears, semen, Pap smear, or cervical, anal, oral, or nasal swabs. On occasion, other relatively non-invasive studies may be indicated. Skin testing with conventional, licensed antigens for assessment of cellular immunity may be performed, and skin lesions may be biopsied or excised. Tumor or other tissue biopsies may be obtained when biopsy or surgery is clinically indicated for other reasons. Otherwise no surgery is performed, and no therapy is administered. Clinical referral to other components of NCI, NIH, or the private sector are made as needed. The biological specimens are frozen or otherwise preserved to be batch tested in current assays or future assays that will be developed. Such laboratory testing is performed either at VEB's own support laboratory, or collaboratively in other NCI, NIH, or extramural laboratories that have the needed expertise for the disease or virus under study.

Occasionally, repeated or more long-term evaluation is required. More often, a single evaluation in the NIH outpatient clinic, or either at a collaborating physician's office or other suitable site in the field, is sufficient. The VEB investigator provides counseling relevant to the virus or disease under study, and about the interim study results. He or she makes appropriate referral if needed (e.g., to the Genetic Epidemiology Branch for genetic counseling). Clinically relevant results and the VEB investigator's interpretation of these results, are provided in writing to the subject's primary caregiver. Confidentiality of the information that is obtained is carefully protected. The results of the study are summarized for publication in the peer review literature.

ELIGIBILITY:
* INCLUSION CRITERIA:

Family or personal medical history of neoplasia of an unusual type, pattern, or number.

Known or suspected factor(s) predisposing to neoplasia, such as environmental exposure (particularly immunological or virological), genetic or congenital factors (Mendelian traits predisposing to neoplasia, birth defects, and chromosomal anomalies), or unusual demographic features.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1996-12-24; Study Completion 2011-10-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States